CLINICAL TRIAL: NCT00342394
Title: Fungicide Exposure Assessment Among Apple and Peach Farmers in the Agricultural Health Study
Brief Title: Fungicide Exposure Assessment Among Apple and Peach Farmers in the Argicultural Health Study
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902049; 02-C-N049
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2013-05-01

CONDITIONS: Pesticides; Occupational Exposure
Keywords: Biological Monitoring; Exposure Determinants; Exposure Validation; Occupational Exposure; Pesticides; Agriculture

SUMMARY:
This protocol describes an exposure assessment study of farmers in North Carolina and Iowa who personally apply the fungicides captan, thiophanate-methyl, and benomyl to apple and peach orchards. The exposure assessment will include environmental measurements as well as biological monitoring data. The biomonitoring data will be based on 24-hour urinary metabolites of the three fungicides selected for study. The study is being done in collaboration with the Argicultural Health Study (AHS), a large prospective health study of licensed private (farmer) and commercial applicators, and the spouses of private applicators. The AHS is sponsored by the National Cancer Institute, the National Institute of Environmental Health Sciences and the Environmental Protection Agency. The study described here will be conducted by the National Institute of Occupational Safety and Health.

In summary, the objectives of this study are 1) to measure actual exposures to the target fungicides using both environmental and biological measures of exposure, 2) to identify and quantify major determinants of exposure, 3) to describe within- and between-worker exposure variability, and 4) to evaluate, to the extent possible, agreement between exposure estimates computed using the AHS exposure algorithms and exposure estimates based on actual measurements.

DETAILED DESCRIPTION:
This protocol describes an exposure assessment study of farmers in North Carolina and Iowa who personally apply the fungicides captan, thiophanate-methyl, and benomyl to apple and peach orchards. The exposure assessment will include environmental measurements as well as biological monitoring data. The biomonitoring data will be based on 24-hour urinary metabolites of the three fungicides selected for study. The study is being done in collaboration with the Agricultural Health Study (AHS), a large prospective health study of licensed private (farmer) and commercial applicators, and the spouses of private applicators. The AHS is sponsored by the National Cancer Institute, the National Institute of Environmental Health Sciences and the Environmental Protection Agency. The study described here will be conducted by the National Institute of Occupational Safety and Health.

Retinal degeneration among applicators in the AHS has been associated with cumulative days of use of five fungicides, including captan and benomyl, which are or have been heavily used in orchards. Minimal monitoring data are available on fungicide exposures among orchard applicators in the U.S. Agent-specific exposure classification in the AHS is based primarily on questionnaire data, supplemented by exposure monitoring data from non-cohort studies in the literature. An algorithm has been developed by AHS to estimate an individual's cumulative exposure using information on duration, frequency and intensity of exposure from questionnaires. The intensity piece of this algorithm identifies factors that either increase or decrease exposure and a "weight" is assigned to each factor to reflect the relative impact of that factor on exposure. Exposure data are need to validate these algorithms, to identify major exposure determinants, and to evaluate the appropriateness of the assigned weights.

Fungicides are applied at regular intervals throughout the spring and summer in orchards. Captan is a frequently applied fungicide that will serve as the primary marker for fungicide exposures in orchards. Participants from the AHS will be selected based on planned use of captan. A benzimidazole fungicide, such as thiophanate-methyl or benomyl, is often applied with captan and exposure to thiophanate-methyl and benomyl will also be monitored. Applicator exposure will be measured using both environmental (air, dermal patch, hand) and biological monitoring methods. Captan is metabolized to tetrahydrophthalimide, which is excreted into the urine. Thiophanate-methyl an benomyl share a common metabolite, methyl (5-hydroxy-1H-benzimidazol-2-yl)-carbamate, which is also excreted into the urine. Dupont is voluntarily withdrawing its benomyl product from the market as of December 31, 2001; however, existing supplies of benomyl may be used in 2002. Due to this "carryover" use of benomyl and the presence of a metabolite in the urine common to thiophanate-methyl, it is prudent to monitor benomyl exposure among participating applicators. A repeated measures design has been proposed to address the likelihood of high within-worker variability for exposure measures.

In summary, the objectives of this study are 1) to measure actual exposures to the target fungicides using both environmental and biological measures of exposure, 2) to identify and quantify major determinants of exposure, 3) to describe within- and between-worker exposure variability, and 4) to evaluate, to the extent possible, agreement between exposure estimates computed using the AHS exposure algorithms and exposure estimates based on actual measurements.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants will be recruited from a sub-sample of the AHS cohort.

To be eligible for this study, AHS participants must:

1. Currently grow apples or peaches and,
2. Plan to personally apply captan during the spring/summer growing season.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2001-11-14; Study Completion 2013-05-01

CONTACTS AND LOCATIONS:
Overall Officials: Michael Alavanja, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institute for Occupational Safety and Health, Atlanta, Georgia, United States

REFERENCES:
- [Background] Carter SD, Laskey JW. Effect of benomyl on reproduction in the male rat. Toxicol Lett. 1982 Apr;11(1-2):87-94. doi: 10.1016/0378-4274(82)90111-4. PMID 7090021
- [Background] Brouwer DH, Brouwer R, De Mik G, Maas CL, van Hemmen JJ. Pesticides in the cultivation of carnations in greenhouses: Part I--Exposure and concomitant health risk. Am Ind Hyg Assoc J. 1992 Sep;53(9):575-81. doi: 10.1080/15298669291360175. PMID 1524032
- [Background] Barnes TB, Verlangieri AJ, Wilson MC. Reproductive toxicity of methyl-1-(butylcarbamoyl)-2-benzimidazole carbamate (benomyl) in male Wistar rats. Toxicology. 1983 Sep;28(1-2):103-15. doi: 10.1016/0300-483x(83)90110-5. PMID 6636195